CLINICAL TRIAL: NCT05307978
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study of Subcutaneously and Intravenously Administered ALXN1910 in Healthy Adult Participants
Brief Title: Safety and Tolerability, Pharmacokinetic, and Pharmacodynamic Study of ALXN1910 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ALXN1910-HV-101
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: ALXN1910; Safety; Pharmacokinetics; Pharmacodynamics; Japanese Descent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Participants will receive a single dose of 5 mg of ALXN1910 IV or Placebo IV.
  Interventions: Drug: ALXN1910; Drug: Placebo
- Cohort 2 (Experimental): Participants will receive a single dose of 15 mg of ALXN1910 SC or Placebo SC.
  Interventions: Drug: ALXN1910; Drug: Placebo
- Cohort 3 (Experimental): Participant will receive a single dose of 15 mg of ALXN1910 IV or Placebo IV.
  Interventions: Drug: ALXN1910; Drug: Placebo
- Cohort 4 (Experimental): Japanese participants will receive a single dose of 15 mg of ALXN1910 SC or Placebo SC.
  Interventions: Drug: ALXN1910; Drug: Placebo
- Cohort 5 (Experimental): Participants will receive a single dose of 45 mg of ALXN1910 SC or Placebo SC.
  Interventions: Drug: ALXN1910; Drug: Placebo
- Cohort 6 (Experimental): Participants will receive a single dose of 135 mg of ALXN1910 SC or Placebo SC.
  Interventions: Drug: ALXN1910; Drug: Placebo

INTERVENTIONS:
Drug: ALXN1910 — Participants will receive a single dose of ALXN1910 IV or ALXN1910 SC according to their assigned cohort.
Drug: Placebo — Participants will receive Placebo IV or Placebo SC according to their assigned cohort.

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of single ascending doses (SADs) of ALXN1910 subcutaneous (SC) and SAD of ALXN1910 intravenous (IV).

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Participants of Japanese descent are defined as: First generation (born to 2 Japanese parents and 4 Japanese grandparents).
* Participants of Japanese descent must be between 20 and 55 years of age.

Exclusion Criteria:

* Current or recurrent disease
* Current or relevant history of physical or psychiatric illness.
* Any other significant disease or disorder that, in the opinion of the Investigator, may put the participant at risk.
* History of significant allergic reaction (eg, anaphylaxis or angioedema) to any product (eg, food, pharmaceutical).
* Female participants who are pregnant or breastfeeding.
* Major surgery or hospitalization within 90 days prior to dosing on Day1.
* History of exposure to asfotase alfa.
* History of allergy or hypersensitivity to excipients of asfotase alfa or ALXN1910 (eg,sodium phosphate, sodium chloride).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Harrow, United Kingdom

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1910-HV-101&attachmentIdentifier=684129f5-6c0c-442c-9ef5-2ca35cf1e4ac&fileName=CSR_synopsis_18_Sep_2023_ALXN1910-HV-101__Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met all the inclusion and none of the exclusion criteria were randomized in 1 site. The study was conducted from 12 Apr 2022 to 07 Feb 2023.
Pre-assignment Details: The screening period was up to 28 days. Informed consent form (ICF) was signed prior to screening procedures. Subjects received study drug in a randomised order. All the study assessments were performed as per the schedule of assessment.
Groups:
- Cohort 1- 5 mg: Participants received a single dose of 5 mg of ALXN1910 IV.
- Cohort 2- 15 mg SC: Participants received a single dose of 15 mg of ALXN1910 SC.
- Cohort 3- 15 mg IV: Participant received a single dose of 15 mg of ALXN1910 IV.
- Japanese Cohort 4- 15 mg SC: Japanese participants received a single dose of 15 mg of ALXN1910 SC.
- Cohort 5- 45 mg: Participants received a single dose of 45 mg of ALXN1910 SC.
- Cohort 6- 135 mg: Participants received a single dose of 135 mg of ALXN1910 SC.
- Pooled Placebo: Participants received a single dose of matching Placebo IV or SC.
Period: Overall Study
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg | Pooled Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12
Completed | 6 | 5 | 6 | 2 | 6 | 6 | 11
Not Completed | 0 | 1 | 0 | 4 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 4 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who receive any amount of study intervention were included in the Safety Set. Participants were analyzed according to the study intervention received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg | Pooled Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 37.7 (9.69) | 33.0 (13.75) | 35.3 (8.89) | 31.8 (7.65) | 30.2 (4.40) | 34.0 (7.85) | 33.6 (6.27) | 33.6 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 2 | 2 | 1 | 6 | 18
  Male | 4 | 3 | 4 | 4 | 4 | 5 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 6 | 5 | 10 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 6 | 0 | 0 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 4 | 3 | 0 | 4 | 4 | 8 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 3 | 0 | 2 | 2 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: The safety and tolerability of ALXN1910 was assessed.
Time Frame: Day 1 (postdose) through Day 75
Population: All participants who received any amount of study intervention were included in the Safety Analysis Set. Participants were analyzed according to the study intervention received.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants
  Any TEAE | 3 | 3 | 4 | 3 | 5 | 4 | 8
  Any Serious TEAE | 0 | 0 | 0 | 0 | 0 | 1 | 0
  TEAE outcome of Death | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AE Leading to Withdrawal of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SAE Leading to Withdrawal of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: The Cmax was assessed as PK parameter of single ascending doses of ALXN1910.
Time Frame: Days 1 through 5 (predose and up to 96 hours postdose), postdose on Days 6, 7, 8, 15, 22, 29, 36, 43, and 75
Population: All treated participants for whom the PK profile of ALXN1910 can be adequately characterized were included in the PK Set. PK analyses were based upon the study intervention received
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
microgram/milliliter (μg/mL) | 1.034 (16.5) | 0.3172 (60.3) | 3.113 (11.5) | 0.3807 (31.8) | 1.230 (32.0) | 4.257 (38.3)

3. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax)
Description: The Tmax was assed as PK parameter of single ascending doses of ALXN1910.
Time Frame: Days 1 through 5 (predose and up to 96 hours postdose), postdose on Days 6, 7, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 2
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour (h) | 0.48 [0.23 to 0.60] | 107.85 [48.01 to 171.50] | 0.52 [0.51 to 0.55] | 108.02 [71.92 to 169.32] | 95.99 [71.89 to 145.03] | 84.14 [48.09 to 142.74]

4. Secondary Outcome: Apparent Terminal Elimination Half Life (t1/2)
Description: The t1/2 was assed as PK parameter of single ascending doses of ALXN1910.
Time Frame: Days 1 through 5 (predose and up to 96 hours postdose), postdose on Days 6, 7, 8, 15, 22, 29, 36, 43, and 75
Population: All treated participants for whom the PK profile of ALXN1910 can be adequately characterized were included in the PK Set. PK analyses were based upon the study intervention received. Here, Number of Participants Analyzed refers to the number of participants available for the specific Outcome measure for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg
Number analyzed (Participants) | 6 | 4 | 6 | 5 | 5 | 6
hour (h) | 166.1 (25.1) | 215.1 (12.2) | 194.9 (19.2) | 207.5 (13.9) | 271.3 (6.0) | 263.5 (18.8)

5. Secondary Outcome: Terminal-phase Elimination Rate Constant (λz)
Description: The λz was assed as PK parameter of single ascending doses of ALXN1910.
Time Frame: Days 1 through 5 (predose and up to 96 hours postdose), postdose on Days 6, 7, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour (1/h)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg
Number analyzed (Participants) | 6 | 4 | 6 | 5 | 5 | 6
1/hour (1/h) | 0.004172 (25.1) | 0.003222 (12.2) | 0.003556 (19.2) | 0.003341 (13.9) | 0.002555 (6.0) | 0.002631 (18.8)

6. Secondary Outcome: AUC From Time Zero to the Last Quantifiable Concentratio (AUCt)
Description: The AUCt was assed as PK parameter of single ascending doses of ALXN1910.
Time Frame: Days 1 through 5 (predose and up to 96 hours postdose), postdose on Days 6, 7, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*μg/mL)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6
hour*microgram/milliliter (h*μg/mL) | 69.52 (23.0) | 102.4 (44.1) | 219.0 (14.2) | 120.9 (30.3) | 484.3 (13.1) | 1606 (20.4)

7. Secondary Outcome: AUC From Time Zero Extrapolated to Infinity (AUC∞)
Description: The AUC∞ was assed as PK parameter of single ascending doses of ALXN1910.
Time Frame: Days 1 through 5 (predose and up to 96 hours postdose), postdose on Days 6, 7, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*μg/mL)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg
Number analyzed (Participants) | 5 | 3 | 6 | 5 | 5 | 6
hour*microgram/milliliter (h*μg/mL) | 89.43 (22.2) | 168.0 (20.3) | 244.5 (13.8) | 157.8 (23.4) | 517.8 (12.4) | 1699 (19.8)

8. Secondary Outcome: AUC From Time Zero to 168h (AUC0-168)
Description: The AUC0-168 was assed as PK parameter of single ascending doses of ALXN1910.
Time Frame: Days 1 through 5 (predose and up to 96 hours postdose), postdose on Days 6, 7, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*μg/mL)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour*microgram/milliliter (h*μg/mL) | 53.06 (14.4) | 40.83 (65.6) | 142.1 (11.6) | 49.73 (35.3) | 161.9 (37.2) | 573.3 (37.9)

9. Secondary Outcome: Percentage of AUC∞ Obtained by Extrapolation Beyond Tlast (%AUCex)
Description: The %AUCex was assed as PK parameter of single ascending doses of ALXN1910.
Time Frame: Days 1 through 5 (predose and up to 96 hours postdose), postdose on Days 6, 7, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage (%) of AUC∞
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg
Number analyzed (Participants) | 6 | 5 | 6 | 5 | 5 | 6
Percentage (%) of AUC∞ | 24.03 (21.1) | 22.89 (73.2) | 10.41 (5.8) | 16.89 (31.8) | 6.418 (12.5) | 5.133 (39.0)

10. Secondary Outcome: Total Body Clearance (for IV Cohorts) or Apparent Clearance (for SC Cohorts) (CL or CL/F)
Description: The CL or CL/F was assed as PK parameter of single ascending doses of ALXN1910.
Time Frame: Days 1 through 5 (predose and up to 96 hours postdose), postdose on Days 6, 7, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg
Number analyzed (Participants) | 5 | 3 | 6 | 5 | 5 | 6
Liter/hour (L/h) | 0.05591 (22.2) | 0.08926 (20.3) | 0.06135 (13.8) | 0.09507 (23.4) | 0.08691 (12.4) | 0.07945 (19.8)

11. Secondary Outcome: Volume of Distribution (for IV Cohorts) or Apparent Volume of Distribution (for SC Cohorts) (Vd or Vd/F)
Description: The Vd or Vd/F was assed as PK parameter of single ascending doses of ALXN1910.
Time Frame: Days 1 through 5 (predose and up to 96 hours postdose), postdose on Days 6, 7, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg
Number analyzed (Participants) | 5 | 3 | 6 | 5 | 5 | 6
Liter (L) | 12.56 (11.2) | 27.12 (29.4) | 17.25 (12.1) | 28.46 (21.0) | 34.02 (11.3) | 30.20 (29.3)

12. Secondary Outcome: Plasma Concentration of Inorganic Pyrophosphate (PPi)
Description: The plasma concentrations of PPi was assesed.
Time Frame: Day 1 (predose), 2, 3, 5, 8, 15, 22, 29, 36, 43, and 75
Population: All treated participants for whom the PD profile of ALXN1910 can be adequately characterized were included in the PD Set. Here, Number Analyzed refers to the number of participants available for the specific Outcome measure for specific timeframe.
Measure: Mean (Standard Deviation); unit: micromole/Liter (umol/L)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
micromole/Liter (umol/L)
  Day 1 | 1.677 (0.6197) | 1.783 (0.5743) | 1.580 (0.2270) | 1.683 (0.2788) | 1.577 (0.2518) | 1.525 (0.2882) | 1.638 (0.3860)
  Day 2 | 1.162 (0.2057) | 1.550 (0.3407) | 0.915 (0.2219) | 1.582 (0.3579) | 1.165 (0.2696) | 0.823 (0.1152) | 1.418 (0.2699)
  Day 3 | 1.152 (0.0719) | 1.303 (0.2728) | 0.950 (0.2134) | 1.405 (0.1733) | 1.093 (0.3075) | 0.778 (0.0694) | 1.408 (0.2405)
  Day 5 | 1.232 (0.1052) | 1.265 (0.2091) | 0.978 (0.2481) | 1.476 (0.4730) | 0.962 (0.2212) | 0.750 (0.750) | 1.509 (0.4246)
  Day 8: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 12
  Day 8 | 1.368 (0.1269) | 1.257 (0.2279) | 1.177 (0.3393) | 1.470 (0.2206) | 0.974 (0.1218) | 0.750 (0) | 1.368 (0.3200)
  Day 15: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 12
  Day 15 | 1.326 (0.0503) | 1.388 (0.1080) | 1.198 (0.1982) | 1.483 (0.2817) | 0.977 (0.1695) | 0.830 (0.1171) | 1.261 (0.1614)
  Day 22: number analyzed (Participants) | 5 | 5 | 6 | 6 | 5 | 6 | 12
  Day 22 | 1.424 (0.1036) | 1.356 (0.1195) | 1.350 (0.2692) | 1.558 (0.1855) | 1.134 (0.1828) | 0.875 (0.1524) | 1.328 (0.1873)
  Day 29: number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 5 | 11
  Day 29 | 1.295 (0.1610) | 1.332 (0.2834) | 1.320 (0.1582) | 1.518 (0.0952) | 1.294 (0.1997) | 1.044 (0.1790) | 1.438 (0.2677)
  Day 36: number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 6 | 12
  Day 36 | 1.417 (0.1845) | 1.455 (0.2036) | 1.412 (0.2226) | 1.516 (0.2192) | 1.308 (0.1760) | 1.180 (0.2347) | 1.413 (0.2283)
  Day 43: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 11
  Day 43 | 1.433 (0.2263) | 1.418 (0.2204) | 1.553 (0.3434) | 1.615 (0.1463) | 1.377 (0.2673) | 1.243 (0.3406) | 1.225 (0.1939)
  Day 75: number analyzed (Participants) | 5 | 4 | 6 | 2 | 6 | 6 | 11
  Day 75 | 1.496 (0.1576) | 1.375 (0.2001) | 1.592 (0.3540) | 1.820 (0.0424) | 1.495 (0.2073) | 1.527 (0.2527) | 1.290 (0.1968)

13. Secondary Outcome: Plasma Concentration of Pyridoxal (PL)
Description: The plasma concentrations of PL was assessed.
Time Frame: Day 1 (predose), 2, 3, 5, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/ml)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
nanogram/milliliter (ng/ml)
  Day 1 | 2.000 (0) | 2.133 (0.3266) | 2.000 (0) | 2.092 (0.2245) | 2.000 (0) | 2.182 (0.3561) | 2.003 (0.0087)
  Day 2: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 12
  Day 2 | 2.000 (0) | 2.078 (0.1919) | 2.000 (0) | 2.000 (0) | 2.000 (0) | 2.395 (0.6874) | 2.000 (0)
  Day 3 | 2.000 (0) | 2.088 (0.1412) | 2.000 (0) | 2.000 (0) | 2.000 (0) | 2.280 (0.5295) | 2.000 (0)
  Day 5 | 2.000 (0) | 2.000 (0) | 2.000 (0) | 2.000 (0) | 2.015 (0.0367) | 2.157 (0.3552) | 2.000 (0)
  Day 8: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 12
  Day 8 | 2.035 (0.0857) | 2.025 (0.0612) | 2.135 (0.3307) | 2.000 (0) | 3.903 (4.6037) | 2.028 (0.0626) | 2.014 (0.0491)
  Day 15: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 12
  Day 15 | 2.108 (0.1855) | 2.000 (0) | 2.000 (0) | 2.850 (1.6067) | 3.877 (4.1356) | 3.430 (2.7195) | 2.183 (0.6319)
  Day 22: number analyzed (Participants) | 5 | 5 | 6 | 6 | 5 | 6 | 12
  Day 22 | 6.230 (8.9909) | 2.000 (0) | 2.017 (0.0408) | 5.042 (5.0662) | 2.140 (0.2706) | 2.725 (1.6564) | 3.904 (4.9090)
  Day 29: number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 5 | 12
  Day 29 | 2.012 (0.0286) | 2.000 (0) | 2.000 (0) | 3.524 (2.8236) | 2.652 (1.4579) | 2.366 (0.7119) | 3.922 (4.4773)
  Day 36: number analyzed (Participants) | 6 | 6 | 6 | 4 | 5 | 6 | 11
  Day 36 | 2.000 (0) | 2.000 (0) | 2.000 (0) | 3.783 (3.5650) | 2.732 (1.5382) | 2.303 (0.3774) | 3.264 (4.1910)
  Day 43: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 11
  Day 43 | 2.000 (0) | 2.000 (0) | 2.000 (0) | 4.368 (4.8417) | 2.797 (1.9368) | 2.052 (0.0816) | 2.119 (0.2683)
  Day 75: number analyzed (Participants) | 5 | 4 | 6 | 2 | 6 | 6 | 11
  Day 75 | 2.000 (0) | 2.000 (0.0700) | 4.033 (4.9806) | 3.305 (1.8455) | 2.498 (0.9561) | 2.580 (0.7991) | 2.525 (1.6742)

14. Secondary Outcome: Plasma Concentration of Pyridoxal 5-Phosphate (PLP)
Description: The plasma concentrations of PLP was assessed.
Time Frame: Day 1 (predose), 2, 3, 5, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/ml)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
nanogram/milliliter (ng/ml)
  Day 1 | 10.187 (4.6534) | 10.332 (3.5662) | 9.817 (4.8904) | 15.883 (5.7614) | 11.503 (6.2856) | 13.940 (4.5167) | 8.789 (3.8742)
  Day 2: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 12
  Day 2 | 7.593 (2.3404) | 9.150 (3.5081) | 6.532 (2.5528) | 11.777 (4.2860) | 10.552 (5.1884) | 6.508 (1.6985) | 8.356 (3.8675)
  Day 3 | 8.148 (2.2653) | 9.398 (3.3232) | 7.110 (2.4781) | 11.487 (4.1591) | 8.182 (3.6379) | 5.737 (1.1692) | 8.753 (4.0128)
  Day 5 | 8.597 (3.5325) | 9.158 (3.4736) | 7.038 (2.0301) | 10.098 (1.6344) | 7.672 (3.2028) | 5.490 (1.2002) | 8.942 (5.0870)
  Day 8: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 12
  Day 8 | 8.753 (3.4828) | 9.443 (2.9710) | 8.190 (5.6565) | 10.572 (3.8381) | 7.562 (2.7438) | 5.270 (0.6037) | 8.960 (4.4173)
  Day 15: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 12
  Day 15 | 10.170 (5.1691) | 8.360 (2.5086) | 8.800 (5.7621) | 18.927 (11.9441) | 9.292 (4.7827) | 10.040 (5.4156) | 10.328 (7.0041)
  Day 22: number analyzed (Participants) | 5 | 5 | 6 | 6 | 5 | 6 | 12
  Day 22 | 13.656 (14.9897) | 8.384 (2.6076) | 9.805 (7.1460) | 30.427 (22.5240) | 10.828 (4.5559) | 10.380 (8.4672) | 20.086 (26.9065)
  Day 29: number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 5 | 12
  Day 29 | 9.722 (2.8996) | 8.758 (4.4855) | 8.610 (2.6303) | 26.354 (24.3632) | 14.880 (10.5484) | 12.682 (7.7458) | 16.309 (21.8318)
  Day 36: number analyzed (Participants) | 6 | 6 | 6 | 4 | 5 | 6 | 11
  Day 36 | 11.115 (4.5799) | 7.932 (2.6500) | 8.118 (3.6145) | 19.608 (19.6025) | 18.514 (12.7452) | 12.318 (3.4330) | 14.191 (15.8284)
  Day 43: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 11
  Day 43 | 10.597 (4.7562) | 8.697 (3.6949) | 8.577 (3.3439) | 22.367 (19.3420) | 16.223 (14.2766) | 9.033 (2.5026) | 10.026 (5.6783)
  Day 75: number analyzed (Participants) | 5 | 4 | 6 | 2 | 6 | 6 | 11
  Day 75 | 12.284 (4.3254) | 9.620 (5.6757) | 10.010 (4.9121) | 17.750 (18.0312) | 14.918 (8.7744) | 15.292 (6.7615) | 13.228 (13.3117)

15. Secondary Outcome: Plasma Concentration of Pyridoxic Acid (PA)
Description: The plasma concentrations of PA was assessed.
Time Frame: Day 1 (predose), 2, 3, 5, 8, 15, 22, 29, 36, 43, and 75
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/ml)
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
nanogram/milliliter (ng/ml)
  Day 1 | 2.613 (0.8986) | 3.088 (0.5566) | 2.988 (1.0540) | 3.590 (1.8724) | 2.750 (0.8456) | 3.797 (1.3833) | 2.798 (0.7626)
  Day 2: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 12
  Day 2 | 2.270 (0.5563) | 2.502 (0.3333) | 2.580 (0.6935) | 3.140 (1.4506) | 2.680 (0.7706) | 2.955 (0.9038) | 2.541 (0.5817)
  Day 3 | 2.273 (0.3469) | 2.828 (0.5980) | 2.558 (0.6787) | 3.240 (1.1469) | 2.463 (0.5376) | 2.828 (0.8422) | 2.751 (0.6523)
  Day 5 | 2.517 (0.4942) | 2.782 (0.5094) | 2.702 (0.5883) | 3.070 (0.9821) | 2.605 (0.5392) | 3.125 (0.3094) | 2.713 (0.5881)
  Day 8: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 12
  Day 8 | 2.680 (1.5016) | 2.797 (1.0017) | 2.733 (0.8122) | 3.497 (1.6013) | 3.012 (1.1908) | 3.054 (0.4078) | 2.939 (0.8534)
  Day 15: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 12
  Day 15 | 2.812 (0.9420) | 3.000 (1.0794) | 2.908 (0.9542) | 5.132 (3.4143) | 3.285 (1.7404) | 6.118 (5.5760) | 2.930 (1.4804)
  Day 22: number analyzed (Participants) | 5 | 5 | 6 | 6 | 5 | 6 | 12
  Day 22 | 10.750 (18.8695) | 2.566 (0.6971) | 3.172 (1.8925) | 10.143 (11.4645) | 3.946 (1.9630) | 4.532 (2.0736) | 5.579 (7.2517)
  Day 29: number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 5 | 12
  Day 29 | 3.453 (1.0153) | 2.575 (0.6291) | 3.070 (1.0623) | 6.922 (7.2945) | 4.576 (3.4900) | 4.482 (2.3754) | 4.553 (4.6084)
  Day 36: number analyzed (Participants) | 6 | 6 | 6 | 4 | 5 | 6 | 11
  Day 36 | 2.833 (1.1429) | 2.657 (0.7266) | 2.563 (1.1121) | 6.185 (7.3577) | 4.236 (2.7877) | 3.950 (1.6757) | 4.557 (4.8259)
  Day 43: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 11
  Day 43 | 2.415 (0.5445) | 2.827 (0.8977) | 3.330 (1.9655) | 8.055 (8.7461) | 4.123 (3.3854) | 3.220 (0.8897) | 3.328 (1.4716)
  Day 75: number analyzed (Participants) | 5 | 4 | 6 | 2 | 6 | 6 | 11
  Day 75 | 3.620 (1.2921) | 2.998 (0.9216) | 2.868 (0.7116) | 6.350 (6.1518) | 3.595 (1.8915) | 4.580 (1.1087) | 3.695 (2.7428)

16. Secondary Outcome: Number of Participants With Positive Treatment-Emergent Antidrug Antibodies (ADAs)
Description: The ADAs of ALXN1910 was assessed as immunogenicity parameter. Treatment-emergent ADA Responses is defined as a positive result in the ADA assay post first dose, when baseline results are negative or missing.
Time Frame: Day 1 (postdose) through Day 75
Population: All randomized/enrolled participants who received at least 1 dose of the study intervention and who after the dose have at least 1 reportable ADA result. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Geometric Mean Ratio (GMR) of Area Under the Curve (AUC∞) Values of Subcutaneous (SC) Versus Intravenous (IV) Serum Concentration of ALXN1910
Description: The absolute bioavailability GMR AUC∞ of ALXN1910 SC was assessed.
Time Frame: Up to Day 75
Population: All treated participants for whom the PK profile of ALXN1910 can be adequately characterized were included in the PK Set. PK analyses were based upon the study intervention received. Here, Number Analyzed refers to the number of participants available for the specific Outcome measure analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: h × μg/mL
Arm/Group | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV
Number analyzed (Participants) | 3 | 6
h × μg/mL | 168.05 [135.38 to 208.59] | 244.51 [209.85 to 284.88]
Statistical Analysis 1: Comparison: Cohort 2- 15 mg SC vs Cohort 3- 15 mg IV; Test type: Superiority; Mixed Models Analysis; A mixed effect model was performed to the ln-transformed PK parameter and the independent variables; Ratio (%) = 68.729, 95% CI 2-sided [52.74 to 89.56]

18. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) in Japanese and Non-Japanese Participants
Description: Quantitative assessment of PK parameter (Cmax) was assessed between Japanese and non-Japanese participants.
Time Frame: Up to Day 75
Population: as for outcome 2
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Cohort 2- 15 mg SC | Japanese Cohort 4- 15 mg SC
Number analyzed (Participants) | 6 | 6
μg/mL | 0.32 [0.21 to 0.48] | 0.38 [0.25 to 0.57]
Statistical Analysis 1: Comparison: Cohort 2- 15 mg SC vs Japanese Cohort 4- 15 mg SC; Test type: Superiority; Mixed Models Analysis; A mixed effect model was performed with ethnicity as fixed effect and participant as random effect; Ratio (%) = 120.043, 95% CI 2-sided [67.20 to 214.43]

19. Secondary Outcome: AUC From Time Zero to the Last Quantifiable Concentration (AUCt) in Japanese and Non-Japanese Participants
Description: Quantitative assessment of PK parameter (AUCt) was assessed between Japanese and non-Japanese participants.
Time Frame: Up to Day 75
Population: as for outcome 2
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: h × μg/mL
Arm/Group | Cohort 2- 15 mg SC | Japanese Cohort 4- 15 mg SC
Number analyzed (Participants) | 6 | 6
h × μg/mL | 102.37 [73.49 to 142.61] | 120.94 [86.82 to 168.48]
Statistical Analysis 1: Comparison: Cohort 2- 15 mg SC vs Japanese Cohort 4- 15 mg SC; Test type: Superiority; Mixed Models Analysis; A mixed effect model was performed with ethnicity as fixed effect and participant as random effect; Ratio (%) = 118.142, 95% CI 2-sided [73.93 to 188.80]

20. Secondary Outcome: AUC From Time Zero Extrapolated to Infinity (AUC∞) in Japanese and Non-Japanese Participants
Description: Quantitative assessment of PK parameter (AUC∞) was assessed between Japanese and non-Japanese participants.
Time Frame: Up to Day 75
Population: as for outcome 17
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: h × μg/mL
Arm/Group | Cohort 2- 15 mg SC | Japanese Cohort 4- 15 mg SC
Number analyzed (Participants) | 3 | 5
h × μg/mL | 168.05 [122.84 to 229.89] | 157.78 [123.78 to 201.12]
Statistical Analysis 1: Comparison: Cohort 2- 15 mg SC vs Japanese Cohort 4- 15 mg SC; Test type: Superiority; Mixed Models Analysis; A mixed effect model was performed with ethnicity as fixed effect and participant as random effect; Ratio (%) = 93.891, 95% CI 2-sided [63.17 to 139.56]

21. Secondary Outcome: Change From Baseline in Inorganic Pyrophosphate Concentration in Japanese and Non-Japanese Participants
Description: Change from baseline in PD parameter Inorganic Pyrophosphate was evaluated over time for Japanese and non-Japanese participants (Cohort 2 versus Cohort 4) on active treatment.
Time Frame: Day 2, 15, 22, 43, and 75
Population: All treated participants for whom the PD profile of ALXN1910 can be adequately characterized were included in the PD Set.
Measure: Least Squares Mean (Standard Error); unit: μmol
Arm/Group | Cohort 2- 15 mg SC | Japanese Cohort 4- 15 mg SC
Number analyzed (Participants) | 6 | 6
μmol
  Day 2 | -0.195 (0.101) | -0.152 (0.101)
  Day 15 | -0.357 (0.101) | -0.251 (0.101)
  Day 22: number analyzed (Participants) | 5 | 6
  Day 22 | -0.355 (0.106) | -0.176 (0.101)
  Day 43 | -0.327 (0.101) | -0.119 (0.101)
  Day 75: number analyzed (Participants) | 4 | 2
  Day 75 | -0.329 (0.114) | -0.015 (0.147)

22. Secondary Outcome: Change From Baseline in Pyridoxal-5-phosphate Concentration in Japanese and Non-Japanese Participants
Description: Change from baseline in PD parameter Pyridoxal-5-phosphate was evaluated over time for Japanese and non-Japanese participants (Cohort 2 versus Cohort 4) on active treatment
Time Frame: Day 2, 15, 22, 43, and 75
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: μmol
Arm/Group | Cohort 2- 15 mg SC | Japanese Cohort 4- 15 mg SC
Number analyzed (Participants) | 6 | 6
μmol
  Day 2 | -0.430 (3.628) | -4.957 (3.659)
  Day 15 | -1.220 (3.628) | 2.193 (3.659)
  Day 22: number analyzed (Participants) | 5 | 6
  Day 22 | -0.412 (3.900) | 13.693 (3.659)
  Day 43 | -0.883 (3.628) | 5.633 (3.659)
  Day 75: number analyzed (Participants) | 4 | 2
  Day 75 | 1.137 (4.269) | 2.839 (5.677)

23. Secondary Outcome: Change From Baseline in Pyridoxal Concentration in Japanese and Non-Japanese Participants
Description: Change from baseline in PD parameter Pyridoxal was evaluated over time for Japanese and non-Japanese participants (Cohort 2 versus Cohort 4) on active treatment.
Time Frame: Day 2, 15, 22, 43, and 75
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Cohort 2- 15 mg SC | Japanese Cohort 4- 15 mg SC
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 2 | -0.093 (0.740) | -0.061 (0.740)
  Day 15 | -0.171 (0.740) | 0.789 (0.740)
  Day 22: number analyzed (Participants) | 5 | 6
  Day 22 | 0.190 (0.795) | 2.981 (0.740)
  Day 43 | -0.171 (0.740) | 2.308 (0.740)
  Day 75: number analyzed (Participants) | 4 | 2
  Day 75 | -0.063 (0.868) | 1.789 (1.174)

24. Secondary Outcome: Change From Baseline in Pyridoxic Acid Concentration in Japanese and Non-Japanese Participants
Description: Change from baseline in PD parameter Pyridoxic Acid was evaluated over time for Japanese and non-Japanese participants (Cohort 2 versus Cohort 4) on active treatment.
Time Frame: Day 2, 15, 22, 43, and 75
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Cohort 2- 15 mg SC | Japanese Cohort 4- 15 mg SC
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 2 | -0.316 (1.263) | -0.725 (1.263)
  Day 15 | 0.182 (1.263) | 1.267 (1.263)
  Day 22: number analyzed (Participants) | 5 | 6
  Day 22 | -0.238 (1.383) | 6.278 (1.263)
  Day 43 | 0.009 (1.263) | 4.190 (1.263)
  Day 75: number analyzed (Participants) | 4 | 2
  Day 75 | 0.189 (1.545) | 4.812 (2.184)

ADVERSE EVENTS:
Time Frame: Day 1 (postdose) through Day 75
Arm/Group | Cohort 1- 5 mg | Cohort 2- 15 mg SC | Cohort 3- 15 mg IV | Japanese Cohort 4- 15 mg SC | Cohort 5- 45 mg | Cohort 6- 135 mg | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 1/6 | 0/12
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 4/6 | 3/6 | 5/6 | 4/6 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1- 5 mg (N=6) | Cohort 2- 15 mg SC (N=6) | Cohort 3- 15 mg IV (N=6) | Japanese Cohort 4- 15 mg SC (N=6) | Cohort 5- 45 mg (N=6) | Cohort 6- 135 mg (N=6) | Pooled Placebo (N=12)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1- 5 mg (N=6) | Cohort 2- 15 mg SC (N=6) | Cohort 3- 15 mg IV (N=6) | Japanese Cohort 4- 15 mg SC (N=6) | Cohort 5- 45 mg (N=6) | Cohort 6- 135 mg (N=6) | Pooled Placebo (N=12)
Catheter site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 3 (4)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral discharge (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
For Outcome measure #12 Plasma Concentration of Inorganic Pyrophosphate (PPi); #13 Plasma Concentration of Pyridoxal (PL); #14 Plasma Concentration of Pyridoxal 5-Phosphate (PLP); 15 Plasma Concentration of Pyridoxic Acid (PA); Cohort 4 Day 75 standard deviation is provided for the posting although standard deviation will not be calculated for less than 3 data points per study's Statistical Analysis Plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT05307978/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT05307978/SAP_001.pdf